CLINICAL TRIAL: NCT05087472
Title: Prevalence of Psychiatric Disorders in the Refugee Population of Turkey
Status: Withdrawn | Type: Observational
Why Stopped: Could not obtain MINI licence
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Suleyman Keles, MD, Psychiatrist, Head of Community Psychiatry Department, Kutahya Health Sciences University
Other Study IDs: 1
Record Dates: First submitted 2021-09-25; First posted 2021-10-21 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are planning to diagnose psychiatric disorders in willing participants from the refugee population in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Having official refugee status in Turkey, willing to participate in the study

Exclusion Criteria:

* Having any disability that prevents answering interviewers' questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients in a primary care clinic who have official refugee status
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Any diagnosed psychiatric disorder using the Mini-International Neuropsychiatric Interview | Through study completion, on average five months
  The Mini-International Neuropsychiatric Interview (M.I.N.I.) is a short structured diagnostic interview designed to screen for DSM-5 and ICD-10 psychiatric disorders. It will be utilized on willing participants from Turkey's refugee population.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No